CLINICAL TRIAL: NCT00284518
Title: Safety and Efficacy Study of Botulinum Toxin Type A to Treat Lower Urinary Symptoms Due to Benign Prostatic Hyperplasia
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Allergan (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 191622-517
Record Dates: First submitted 2006-01-31; First posted 2006-02-01 (Estimated); Results first posted 2012-12-17 (Estimated); Last update posted 2012-12-17 (Estimated); Status verified 2012-11

CONDITIONS: Benign Prostatic Hyperplasia
MeSH Terms: conditions — Prostatic Hyperplasia | interventions — Botulinum Toxins, Type A; Saline Solution

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- botulinum toxin Type A 300 U (Experimental): Botulinum toxin Type A 300 U transperineal or transrectal injection on Day 1.
  Interventions: Biological: botulinum toxin Type A
- botulinum toxin Type A 200 U (Experimental): Botulinum toxin Type A 200 U transperineal or transrectal injection on Day 1.
  Interventions: Biological: botulinum toxin Type A
- botulinum toxin Type A 100 U (Experimental): Botulinum toxin Type A 100 U transperineal or transrectal injection on Day 1.
  Interventions: Biological: botulinum toxin Type A
- Placebo (Normal Saline) (Placebo Comparator): Placebo (Normal Saline) transperineal or transrectal injection on Day 1.
  Interventions: Drug: normal saline

INTERVENTIONS:
Biological: botulinum toxin Type A — Botulinum toxin Type A 300 U, 200 U or 100 U transperineal or transrectal injection on Day 1.
  Other Names: BOTOX®
  Arms: botulinum toxin Type A 100 U; botulinum toxin Type A 200 U; botulinum toxin Type A 300 U
Drug: normal saline — Normal Saline (Placebo) transperineal or transrectal injection on Day 1.
  Arms: Placebo (Normal Saline)

SUMMARY:
The purpose of this study was to determine the safety and effectiveness of different doses of botulinum toxin Type A in treating lower urinary tract symptoms due to benign prostatic hyperplasia.

ELIGIBILITY:
Inclusion Criteria:

* Lower urinary tract symptoms due to benign prostatic hyperplasia
* Enlarged prostate volume by rectal ultrasound

Exclusion Criteria:

* Previous prostate surgery
* Previous or current diagnosis of prostate cancer
* Use of other medications for the treatment of prostatic hyperplasia
* Urinary tract infection

Min Age: 50 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 380 (Actual)
Dates: Start 2005-12; Primary Completion 2009-05 (Actual); Study Completion 2010-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Allergan
Locations (11):
- Murdoch, Australia
- Vienna, Austria
- Victoria, British Columbia, Canada
- Olomouc, Czechia
- Paris, France
- Braunschweig, Germany
- Perugia, Italy
- Martin, Slovakia
- Seoul, South Korea
- Taipei, Taiwan
- London, United Kingdom

REFERENCES:
- [Derived] Marberger M, Chartier-Kastler E, Egerdie B, Lee KS, Grosse J, Bugarin D, Zhou J, Patel A, Haag-Molkenteller C. A randomized double-blind placebo-controlled phase 2 dose-ranging study of onabotulinumtoxinA in men with benign prostatic hyperplasia. Eur Urol. 2013 Mar;63(3):496-503. doi: 10.1016/j.eururo.2012.10.005. Epub 2012 Oct 12. PMID 23098762

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Botulinum Toxin Type A 300 U | Botulinum Toxin Type A 200 U | Botulinum Toxin Type A 100 U | Placebo (Normal Saline)
Started | 97 | 94 | 95 | 94
Completed | 71 | 66 | 67 | 61
Not Completed | 26 | 28 | 28 | 33

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Botulinum Toxin Type A 300 U | Botulinum Toxin Type A 200 U | Botulinum Toxin Type A 100 U | Placebo (Normal Saline) | Total
Number analyzed (Participants) | 97 | 94 | 95 | 94 | 380
Age, Customized [Number; unit: Participants]
  45 to 65 Years | 48 | 46 | 56 | 44 | 194
  >65 Years | 49 | 48 | 39 | 50 | 186
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 0 | 0 | 0 | 0
  Male | 97 | 94 | 95 | 94 | 380

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in International Prostate Symptom Score (IPSS) at Week 12
Description: The International Prostate Symptom Score is a disease-specific outcome measure based on the American Urological Association Symptom Index. The questionnaire consists of seven items. The patient evaluates their urinary symptoms (incomplete emptying, frequency, hesitancy, urgency, weak stream, straining, and nocturia) during the previous 4 weeks. The total symptom score can range from 0 (no symptoms) to 35 (most severe symptoms). A negative change from baseline indicates improvement.
Time Frame: Baseline, Week 12
Population: Participants from the intent-to-treat population (includes all randomized participants) with data available for analyses at the given time-point.
Measure: Mean (Standard Deviation); unit: Score on a scale
Arm/Group | Botulinum Toxin Type A 300 U | Botulinum Toxin Type A 200 U | Botulinum Toxin Type A 100 U | Placebo (Normal Saline)
Number analyzed (Participants) | 89 | 91 | 94 | 92
Score on a scale
  Baseline | 21.3 (6.03) | 20.2 (5.80) | 21.5 (5.42) | 20.7 (5.44)
  Change from baseline at Week 12 (N=86,89,93,90) | -5.6 (7.73) | -6.3 (7.13) | -6.6 (6.87) | -5.5 (6.33)

2. Secondary Outcome: Change From Baseline in International Prostate Symptom Score (IPSS) at Week 72
Description: as for outcome 1
Time Frame: Baseline, Week 72
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Score on a scale
Arm/Group | Botulinum Toxin Type A 300 U | Botulinum Toxin Type A 200 U | Botulinum Toxin Type A 100 U | Placebo (Normal Saline)
Number analyzed (Participants) | 89 | 91 | 94 | 92
Score on a scale
  Baseline | 21.3 (6.03) | 20.2 (5.80) | 21.5 (5.42) | 20.7 (5.44)
  Change from baseline at Week 72 (N=64,61,66,58) | -5.0 (6.50) | -4.1 (6.40) | -4.7 (7.15) | -4.3 (7.15)

3. Secondary Outcome: Change From Baseline in Peak Urine Flow Rate
Description: Urinary flow was determined by uroflowmetry at baseline and various time-points during the study. An increase from baseline indicates improvement.
Time Frame: Baseline, Week 12, Week 72
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: milliliters (mL)/second
Arm/Group | Botulinum Toxin Type A 300 U | Botulinum Toxin Type A 200 U | Botulinum Toxin Type A 100 U | Placebo (Normal Saline)
Number analyzed (Participants) | 95 | 89 | 93 | 91
milliliters (mL)/second
  Baseline | 10.4 (2.70) | 10.6 (2.83) | 9.6 (2.57) | 10.1 (2.82)
  Change from baseline to Week 12 (N=81,80,86,77) | 1.8 (4.65) | 2.0 (4.98) | 2.7 (5.21) | 2.8 (4.74)
  Change from baseline to Week 72 (N=59,56,64,53) | 2.0 (4.67) | 2.4 (5.18) | 2.0 (4.07) | 2.3 (4.31)

4. Secondary Outcome: Change From Baseline in Total Prostate Volume
Description: Measurement of the prostate volume was performed via transrectal ultrasound at baseline and various time-points during the study. The prostate gland was scanned and the volume was calculated using the formula: Volume (mL) = length × width × height × 0.523. A negative change from baseline indicates improvement.
Time Frame: Baseline, Week 12, Week 72
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: milliliter (mL)
Arm/Group | Botulinum Toxin Type A 300 U | Botulinum Toxin Type A 200 U | Botulinum Toxin Type A 100 U | Placebo (Normal Saline)
Number analyzed (Participants) | 96 | 91 | 92 | 91
milliliter (mL)
  Baseline | 48.78 (16.800) | 48.40 (16.325) | 47.54 (16.917) | 47.23 (14.867)
  Change from baseline at Week 12 (N=86,84,88,82) | -3.40 (10.046) | -3.65 (9.255) | -3.54 (9.823) | -4.59 (8.392)
  Change from baseline at Week 72 (N=65,60,67,57) | -3.58 (9.773) | -2.82 (11.194) | -1.77 (10.714) | -2.69 (10.875)

5. Secondary Outcome: Change From Baseline in Transitional Zone Prostate Volume
Description: Measurement of the transitional zone prostate volume was performed via transrectal ultrasound at baseline and various time-points during the study. The prostate gland was scanned and the volume was calculated using the formula: Volume (mL) = length × width × height × 0.523. A negative change from baseline indicates improvement.
Time Frame: Baseline, Week 12, Week 72
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: milliliters (mL)
Arm/Group | Botulinum Toxin Type A 300 U | Botulinum Toxin Type A 200 U | Botulinum Toxin Type A 100 U | Placebo (Normal Saline)
Number analyzed (Participants) | 94 | 89 | 90 | 87
milliliters (mL)
  Baseline | 20.78 (14.657) | 21.75 (12.931) | 21.00 (14.188) | 20.73 (13.210)
  Change from baseline at Week 12 (N=83,82,86,79) | -0.23 (6.516) | -0.76 (8.085) | -0.02 (8.445) | -0.27 (6.551)
  Change from baseline at Week 72 (N=64,59,65,55) | 0.19 (7.655) | -0.94 (8.119) | -0.35 (8.808) | -1.35 (6.801)

6. Secondary Outcome: Change From Baseline in Post-Void Residual
Description: Post-void residual urine volume was assessed by bladder scan or ultrasound on all participants at baseline and various time-points during the study. After voiding, any residual urine volume in the bladder was measured. A negative change from baseline indicates improvement.
Time Frame: Baseline, Week 2, Week 12, Week 72
Population: Participants from the safety population (includes all randomized and treated participants) with data available for analyses at the given time-point.
Measure: Mean (Standard Deviation); unit: milliliters (mL)
Arm/Group | Botulinum Toxin Type A 300 U | Botulinum Toxin Type A 200 U | Botulinum Toxin Type A 100 U | Placebo (Normal Saline)
Number analyzed (Participants) | 92 | 89 | 89 | 91
milliliters (mL)
  Baseline | 73.0 (57.07) | 69.7 (54.93) | 66.1 (55.59) | 64.3 (51.89)
  Change from baseline at Week 2 (N=76,82,80,78) | 5.4 (64.06) | 10.9 (88.62) | -1.4 (65.01) | 1.6 (61.03)
  Change from baseline at Week 12 (N=88,84,89,82) | 7.5 (78.18) | 9.0 (81.23) | -1.4 (62.82) | 3.2 (57.92)
  Change from baseline at Week 72 (N=66,60,65,60) | 10.9 (73.27) | -12.4 (54.31) | 14.0 (75.97) | 6.0 (69.79)

7. Other Pre Specified Outcome: Change From Baseline in the International Index of Erectile Function (IIEF) Questionnaire Erectile Function Domain
Description: The IIEF is a 15-item questionnaire filled out by the patient to assess erectile function over the past 4 weeks that contains five domains. The score for the erectile function domain is the sum of scores for Questions 1, 2, 3, 4, 5 and 15 for a total possible score of 1 to 30. A higher score indicates a better outcome. A positive change from baseline indicates improvement.
Time Frame: Baseline, Week 12, Week 72
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Score on a scale
Arm/Group | Botulinum Toxin Type A 300 U | Botulinum Toxin Type A 200 U | Botulinum Toxin Type A 100 U | Placebo (Normal Saline)
Number analyzed (Participants) | 86 | 79 | 84 | 87
Score on a scale
  Baseline | 15.4 (10.20) | 14.6 (10.7) | 17.2 (10.19) | 16.7 (10.29)
  Change from baseline at Week 12 (N=80,72,83,79) | 0.1 (6.66) | -0.2 (5.54) | -0.9 (6.93) | 1.3 (7.86)
  Change from baseline at Week 72 (N=61,54,61,58) | 0.8 (7.17) | 0.5 (4.56) | -1.5 (7.34) | -0.9 (7.95)

8. Post Hoc Outcome: Change From Baseline in IPSS at Week 12 in Patients Previously Treated With Alpha-blockers
Description: The International Prostate Symptom Score (IPSS) is a disease-specific outcome measure based on the American Urological Association Symptom Index. The questionnaire consists of seven items. The patient evaluates their urinary symptoms (incomplete emptying, frequency, hesitancy, urgency, weak stream, straining, and nocturia) during the previous 4 weeks. The total symptom score can range from 0 (no symptoms) to 35 (most severe symptoms). A negative change from baseline indicates improvement.
Time Frame: Baseline, Week 12
Population: Participants from the Intent-to-treat population previously treated with alpha-blockers with data available for analyses.
Measure: Mean (Standard Deviation); unit: Score on a scale
Arm/Group | Botulinum Toxin Type A 300 U | Botulinum Toxin Type A 200 U | Botulinum Toxin Type A 100 U | Placebo (Normal Saline)
Number analyzed (Participants) | 44 | 35 | 52 | 43
Score on a scale
  Baseline | 21.3 (6.20) | 19.6 (6.15) | 21.9 (5.65) | 20.4 (5.32)
  Change from baseline at Week 12 (N=44,35,52,42) | -5.1 (7.76) | -6.6 (5.91) | -5.4 (5.17) | -3.5 (6.12)

ADVERSE EVENTS:
Description: Safety population was used to calculate the number of participants at risk for Serious Adverse Events and Adverse Events and was defined as all randomized and treated participants.
Arm/Group | Botulinum Toxin Type A 300 U | Botulinum Toxin Type A 200 U | Botulinum Toxin Type A 100 U | Placebo (Normal Saline)
Serious Adverse Events (participants affected / at risk) | 9/94 | 16/93 | 10/94 | 11/92
Other Adverse Events (participants affected / at risk) | 41/94 | 46/93 | 53/94 | 55/92
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Botulinum Toxin Type A 300 U (N=94) | Botulinum Toxin Type A 200 U (N=93) | Botulinum Toxin Type A 100 U (N=94) | Placebo (Normal Saline) (N=92)
Angina pectoris (Cardiac disorders) | 0 | 2 | 0 | 0
Angina unstable (Cardiac disorders) | 0 | 1 | 0 | 0
Myocardial infarction (Cardiac disorders) | 0 | 1 | 0 | 0
Acute coronary syndrome (Cardiac disorders) | 0 | 0 | 2 | 0
Blindness unilateral (Eye disorders) | 0 | 0 | 1 | 0
Retinal artery thrombosis (Eye disorders) | 0 | 0 | 1 | 0
Corneal degeneration (Eye disorders) | 0 | 0 | 0 | 1
Gastritis (Gastrointestinal disorders) | 0 | 1 | 0 | 0
Intestinal obstruction (Gastrointestinal disorders) | 0 | 1 | 0 | 0
Inguinal hernia (Gastrointestinal disorders) | 0 | 0 | 1 | 0
Accidental death (General disorders) | 0 | 2 | 0 | 0
Non-cardiac chest pain (General disorders) | 0 | 0 | 1 | 0
Cholecystitis acute (Hepatobiliary disorders) | 0 | 1 | 0 | 0
Cholelithiasis (Hepatobiliary disorders) | 0 | 1 | 0 | 0
Herpes zoster (Infections and infestations) | 0 | 1 | 0 | 0
Bacterial prostatitis (Infections and infestations) | 0 | 0 | 0 | 1
Cellulitis (Infections and infestations) | 0 | 0 | 0 | 1
Femur fracture (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0
Prostatic specific antigen increased (Investigations) | 1 | 0 | 0 | 0
Arthritis (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0
Intervertebral disc protrusion (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 2
Prostate cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0 | 0
Renal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0 | 1
Renal cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0 | 0
Metastatic neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1 | 0
Basal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 1
Gastric adenoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 1
Gastric cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 1
Hypoaesthesia (Nervous system disorders) | 1 | 0 | 0 | 0
Carotid artery stenosis (Nervous system disorders) | 0 | 0 | 0 | 1
Alcoholism (Psychiatric disorders) | 0 | 1 | 0 | 0
Anxiety (Psychiatric disorders) | 0 | 0 | 1 | 0
Calculus bladder (Renal and urinary disorders) | 2 | 0 | 0 | 0
Urinary retention (Renal and urinary disorders) | 1 | 0 | 1 | 0
Nephrolithiasis (Renal and urinary disorders) | 1 | 0 | 0 | 0
Calculus ureteric (Renal and urinary disorders) | 0 | 0 | 1 | 0
Hydronephrosis (Renal and urinary disorders) | 0 | 0 | 1 | 0
Prostatitis (Reproductive system and breast disorders) | 1 | 2 | 1 | 0
Benign prostatic hyperplasia (Reproductive system and breast disorders) | 0 | 1 | 0 | 1
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0
Hypertensive crisis (Vascular disorders) | 0 | 1 | 0 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Botulinum Toxin Type A 300 U (N=94) | Botulinum Toxin Type A 200 U (N=93) | Botulinum Toxin Type A 100 U (N=94) | Placebo (Normal Saline) (N=92)
Urinary tract infection (Infections and infestations) | 6 | 1 | 4 | 3
Nasopharyngitis (Infections and infestations) | 5 | 6 | 5 | 5
Prostatic specific antigen increase (Investigations) | 5 | 5 | 3 | 5
Back pain (Musculoskeletal and connective tissue disorders) | 1 | 5 | 2 | 3
Renal cyst (Renal and urinary disorders) | 7 | 2 | 7 | 3
Haematuria (Renal and urinary disorders) | 4 | 7 | 8 | 8
Urinary retention (Renal and urinary disorders) | 2 | 2 | 5 | 3
Dysuria (Renal and urinary disorders) | 2 | 5 | 4 | 3
Micturition urgency (Renal and urinary disorders) | 1 | 3 | 5 | 6
Pollakiuria (Renal and urinary disorders) | 1 | 2 | 2 | 5
Haematospermia (Reproductive system and breast disorders) | 2 | 6 | 5 | 7
Hypertension (Vascular disorders) | 5 | 2 | 3 | 4

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
A disclosure restriction on the PI is that the sponsor can review results communications prior to public release and can embargo communications regarding trial results for a period that is less than or equal to 90 days from the time submitted to the sponsor for review. The sponsor cannot require changes to the communication and cannot extend the embargo.